CLINICAL TRIAL: NCT06179303
Title: A Phase II Trial to Evaluate Functional Imaging in Prediction of Response to Abemaciclib for Advanced Hormone Receptor-Positive, HER2-Negative Breast Cancer
Brief Title: Functional Imaging in Prediction of Response to Abemaciclib for Advanced Hormone Receptor-Positive, HER2-Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122019; NCI-2022-06409 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020029 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-12-08; First posted 2023-12-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Unresectable HER2-Negative Breast Carcinoma; Locally Advanced Unresectable Hormone Receptor-Positive Breast Carcinoma; Metastatic HER2-Negative Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: interventions — abemaciclib; Anastrozole; Specimen Handling; X-Rays; exemestane; Fluorodeoxyglucose F18; Fulvestrant; Gonadotropin-Releasing Hormone; Letrozole; Magnetic Resonance Spectroscopy; Tamoxifen; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FFNP-PET/CT, estradiol, abemaciclib, ET) (Experimental): Patients receive FFNP IV and undergo PET/CT imaging at baseline. Patients then receive estradiol orally Q8H over a 24-hour period, followed again by FFNP IV and PET/CT imaging. Patients then receive abemaciclib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive ET of the treating physician choice. Patients also receive FDG IV and undergo PET/CT imaging at baseline, with additional diagnostic imaging for tumor assessment every 3 cycles, and undergo blood sample collection throughout the study.
  Interventions: Drug: Abemaciclib; Drug: Anastrozole; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Diagnostic Imaging Testing; Drug: Exemestane; Other: Fludeoxyglucose F-18; Drug: Fluorine F 18 Fluoro Furanyl Norprogesterone; Drug: Fulvestrant; Biological: Gonadotropin-releasing Hormone Analog; Drug: Letrozole; Procedure: Positron Emission Tomography; Drug: Tamoxifen; Drug: Therapeutic Estradiol

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Diagnostic Imaging Testing — Undergo clinical imaging for tumor assessment
  Other Names: Diagnostic Imaging; Medical Imaging
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Fluorine F 18 Fluoro Furanyl Norprogesterone — Given IV
  Other Names: [18F]FFNP
Drug: Fulvestrant — Given IM injection
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Biological: Gonadotropin-releasing Hormone Analog — Given GnRH analog
  Other Names: GnRH Agonist; GnRH Analog; Gonadotropin-Releasing Hormone Agonist; Gonadotropin-Releasing Hormone Analogue; LH-RH agonist; LH-RH Analogs; LHRH Agonist; luteinizing hormone-releasing hormone agonist; Luteinizing Hormone-Releasing Hormone Analog
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara; Fempro
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Tamoxifen — Given PO
  Other Names: TMX
Drug: Therapeutic Estradiol — Given PO
  Other Names: 17 Beta-Estradiol; Aquadiol; Climara; Dimenformon; Diogyn; Diogynets; Estrace; ESTRADIOL; Estraldine; Oestradiol; Ovocylin; Progynon; Vagifem

SUMMARY:
This phase II trial tests the accuracy of functional imaging (FFNP)-positron emission tomography (PET)/computed tomography (CT) to predict response to abemaciclib plus endocrine therapy. Abemaciclib is a drug used to treat certain types of hormone receptor positive (HR+), HER2 negative breast cancer. Abemaciclib blocks certain proteins, which may help keep tumor cells from growing. Endocrine therapy adds, blocks, or removes hormones that can cause cancer to grow. FFNP PET imaging is a form of x-ray that uses FFNP as an imaging agent that may provide more precise information about the location of tumors that "light up" with FFNP than a PET scan alone can provide.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive FFNP intravenously (IV) and undergo PET/CT imaging at baseline. Patients then receive estradiol orally every 8 hours (Q8H) over a 24-hour period, followed again by FFNP IV and PET/CT imaging. Patients then receive abemaciclib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive endocrine therapy (ET) of the treating physician choice. Patients also receive FDG IV and undergo PET/CT imaging at baseline, with additional diagnostic imaging for tumor assessment every 3 cycles, and undergo blood sample collection throughout the study.

After study completion of study, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with metastatic or locally advanced unresectable breast cancer
* Histologically confirmed ER+ / HER2-negative, breast cancer who is a candidate for endocrine therapy with pathology from the primary tumor or metastatic/recurrent site. Based on American Society of Clinical Oncology/College of American Pathologists (ASCO CAP) Guidelines: ER+: >= 1% of tumor cell nuclei to be immunoreactive. HER2-negative: HER2 of 0, 1+ by immunohistochemistry (IHC) or negative by fluorescence in situ hybridization (FISH).

  * In the case of bone biopsy which could yield false negative ER or PR status in patients with historically HR+ disease, a patient may be eligible if the treating physician and the study chair both agree that the patient is a candidate for further endocrine therapy (ET) based treatment.
  * Note that baseline PR status by IHC does not influence results of deltaFFNP-PET imaging.
* If premenopausal, the patient has to be treated with GnRH agonist for at least 6 weeks prior to FFNP-PET.
* Disease must be present in at least one non-liver site and measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and be 1.5 cm or greater in longest dimension OR disease can be non-measurable but must be 1.5 cm in longest dimension on functional imaging (fluorodeoxyglucose [FDG]-PET/computed tomography [CT] preferred).
* No limits to prior lines of endocrine therapy in the metastatic setting including synergistic targeted therapy such as CDK4/6 inhibitors (other than Abemaciclib), PI3K inhibitor, mTOR inhibitor, etc. One line of prior cytotoxic chemotherapy in the metastatic setting is allowed. Washout from prior systemic anti-cancer therapy of at least 2 weeks from chemotherapy or radiation, 2 weeks or 5 half lives (whichever is longer) from oral selective estrogen receptor degrader (SERD), 8 weeks from oral selective estrogen receptor modulator (SERM), and 16 weeks from intramuscular SERD (Fulvestrant) is required. Recovery of adverse events from the last therapy to grade 1 except alopecia. Patients may continue luteinizing hormone-releasing hormone (LHRH) agonist to remain post-menopausal without a need for washout
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* At least 18 years of age
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN).

  * In case of known Gilbert's syndrome, < 2 x ULN is allowed
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) /alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) =< 2.5x institutional ULN, or =< 5 x ULN for subjects with documented metastatic disease to the liver
* eGFR (estimated glomerular filtration rate) ≥ 30 mL/min
* Women of childbearing potential must agree to use adequate contraception (barrier method of birth control, abstinence) prior to study entry and for the duration of study participation
* Ability to understand and willingness to sign an institutional review board (IRB)-approved written informed consent document (or that of legally authorizes representative, if applicable)
* Consent to access archival tumor specimens for clinical sequencing data of tumor tissue and blood

Exclusion Criteria:

* Prior abemaciclib in the metastatic setting or within 2 years of completion of adjuvant abemaciclib
* Hepatic-only metastatic disease
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease
* Currently receiving any other investigational agents
* Untreated/unstable brain metastases. Patients with treated/stable brain metastases, defines as patients who have received prior therapy for their brain metastases and whose central nervous system (CNS) disease is radiographically stable at study entry, are eligible
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to FFNP, abemaciclib, or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Pregnant and/or breastfeeding women of childbearing potential must have a negative pregnancy test within 14 days of study entry. Male participants and female participants of childbearing potential must utilize adequate contraceptive methods throughout study treatment and for at least 30 days after the last dose of study medications
* Patients with human immunodeficiency virus (HIV) are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective antiretroviral therapy (ART) according to Department of Health and Human Services (DHHS) treatment guidelines is recommended

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Response to abemaciclib + endocrine therapy | Up to 2 years
  Non-responding: progression within 24 weeks by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death due to disease within 24 weeks or stable disease but lasting less than 24 weeks. Responding: defined as complete response (CR), partial response (PR) or stable disease lasting >= 24 weeks. Quantitative deltaFFNP will be summarized by descriptive statistics (mean, median, standard deviation [SD], etc.) and tested against 0 by Wilcoxon signed rank test or paired t-test as appropriate, overall and by response. The dichotomized deltaFFNP will be summarized by count and percentages, overall and by response.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Defined by RECIST 1.1
Progression free survival rate (PFS) | Up to 2 years
  Defined from date on study to date of progression or date of death or date of last clinical follow up with imaging evidence showing no progression if a patient did not progress or die, whichever the earliest. PFS events include progression and death.
Overall survival rate (OS) | Up to 2 years
  Defined from date on study to date of death or last follow up if a patient is still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No